CLINICAL TRIAL: NCT05731492
Title: A Multicenter, Open-label, Single-arm Study to Assess the Pharmacokinetics and Safety of Macitentan in Children Aged 1 Month to <2 Years With Pulmonary Arterial Hypertension
Brief Title: A Study of Macitentan in Children Below 2 Years of Age
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR109286; 2022-002754-74 (EudraCT Number); 67896062PAH1013 (Other: Actelion Pharmaceuticals Ltd)
Record Dates: First submitted 2023-02-09; First posted 2023-02-16 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Arterial Hypertension, Pulmonary
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label Core Treatment Period: Macitentan (Experimental): Participants will receive macitentan as a monotherapy or add-on to an existing therapy daily for 24 weeks during core treatment period. Optional treatment extension period of up to 1 year for those participants who completed the core treatment period.
  Interventions: Drug: Macitentan

INTERVENTIONS:
Drug: Macitentan — Macitentan will be administered orally.
  Other Names: JNJ-67896062; ACT-064922

SUMMARY:
The purpose of this study is to learn what happens to macitentan and its active metabolite (aprocitentan) in the body of children aged between 1 month and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary arterial hypertension (PAH): 1) including participants with Down syndrome. Diagnosis must have been confirmed by (historical, any time before screening) right heart catheterization mean pulmonary arterial pressure (mPAP) greater than or equal to (>=) 25 millimeter of mercury (mmHg), pulmonary arterial wedge pressure (PAWP) less than or equal to (=<)15 mmHg, pulmonary vascular resistance index greater than (>) 3 Wood units * meter square (m^2) where in the absence of pulmonary vein obstruction and/or significant lung disease PAWP can be replaced left atrium pressure or left ventricular end diastolic pressure (in the absence of mitral stenosis) assessed by heart catheterization. a) Idiopathic PAH, or b) Heritable PAH, or c) PAH associated with congenital heart disease: i) Eisenmenger syndrome (Qp/Qs less than (<) 1.5 and saturation of peripheral oxygen ≤ 90 percent (%) measured by pulse oximetry at room air), or ii) Inoperable open left-to-right shunts (with a Pulmonary vascular resistance [PVR] > 8 WU and Qp/Qs <2), or iii) Co-incidental shunt (that is, not explaining hemodynamically the presence of PAH), or iv) Post-operative PAH (persisting/recurring/developing ≥ 6 months after repair of shunt), or d) Drug or toxin induced PAH, or e) PAH associated with Human immunodeficiency viruses (HIV)
* World Health Organization Functional Class (WHO FC) I, II, or III
* PAH-specific treatment-naive participants or participants on PAH specific monotherapy or combination of 2 therapies. Use of macitentan before or during screening is allowed
* Body weight of greater than or equal to (>=) 3.5 kilogram (kg)
* Parent(s) (preferably both if available or as per local requirements) or participant's legally designated representative must sign an informed consent form (ICF) indicating that they understand the purpose of, and procedures required for, the study and is/are willing to allow the child to participate in the study

Exclusion Criteria:

* PAH due to portal hypertension, schistosomiasis, pulmonary veno-occlusive disease and/or pulmonary capillary hemangiomatosis
* Persistent pulmonary hypertension of the newborn
* The following congenital cardiac abnormalities: a) Cyanotic congenital cardiac lesions such as transposition of the great arteries, truncus arteriosus, pulmonary atresia with ventricular septal defect, unless operatively repaired and with no residual shunt. b) Univentricular heart and/or participants with Fontan-palliation
* Pulmonary hypertension due to lung disease
* Known diagnosis of bronchopulmonary dysplasia

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-03-14 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Trough Concentration of Macitentan and its Active Metabolite Aprocitentan at Week 4 in Steady-State | Predose (at Week 4)
  Trough concentration of macitentan and its active metabolite aprocitentan at week 4 in steady-state will be reported.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 1.5 years
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.
Number of Participants with Serious Adverse Events (SAEs) | Up to 1.5 years
  A SAE is any AE that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect and is a suspected transmission of any infectious agent via a medicinal product, is medically important.
Number of Participants with AEs Leading to Premature Discontinuation of Macitentan | Up to 1.5 years
  Number of participants with AEs Leading to premature discontinuation of macitentan will be reported.
Number of Participants with Adverse Event of Special Interests (AESIs) | Up to 1.5 years
  Number of participants with AESI will be reported. AEs considered to be of special interest are as hypotension, edema/fluid retention, hemoglobin decrease/anemia, liver events.
Number of Participants with Clinical Laboratory Abnormalities | Up to 1.5 years
  Number of participants with clinical laboratory abnormalities (serum, chemistry and hematology) will be reported.
Number of Participants with Change from Baseline in Clinical laboratory Values. | Up to 1.5 years
  Number of participants with change from baseline in clinical laboratory values will be reported.
Change from Baseline in Blood Pressure | Up to 1.5 years
  Change from baseline in blood pressure will be reported.
Change From Baseline in Heart Rate | Up to 1.5 years
  Change from baseline in heart rate will be reported.
Change From Baseline in Body Weight | Up to 1.5 years
  Change from baseline in body weight will be reported.
Change From Baseline in Length | Up to 1.5 years
  Change from baseline in length will be reported.
Change from Baseline in Height | Up to 1.5 years
  Change from baseline in height will be reported.
Plasma Concentration of Macitentan and its Active Metabolite (Aprocitentan) for Macitentan Naive Participants | At 2, 5, and 24 hours after the first dose of macitentan on Day 1
  Plasma concentrations of macitentan and its active metabolite (aprocitentan) after the first dose of macitentan for macitentan naive participants will be reported.
Trough Concentrations of Macitentan and its Active Metabolite Aprocitentan at Week 8 in Steady-State Conditions | Predose (at Week 8)
  Trough concentrations of macitentan and its active metabolite aprocitentan at week 8 in steady-state conditions will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Pharmaceuticals Ltd Clinical Trial, Study Director — Actelion
Locations (4):
- Germany (2):
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Universitatsmedizin Gottingen, Göttingen
- Poland (2):
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw
  - Wojewodzki Szpital Specjalistyczny We Wroclawiu, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency